CLINICAL TRIAL: NCT03909867
Title: Detection of the Human Aerosolization Patterns of Respiratory Syncytial Virus
Brief Title: Emission Patterns of Respiratory Syncytial Virus
Status: Terminated | Type: Observational
Why Stopped: The emergence of SARS-CoV-2 required hold of recruitment
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00056852
Record Dates: First submitted 2019-04-03; First posted 2019-04-10 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-07

CONDITIONS: RSV Infection; Aerosol Disease
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — One nasopharyngeal swab sample from each participant will be used to confirm RSV infection and determine the amount of the pathogen carried by the individual.
  One-time air samples will be collected using six-stage Andersen air sampling devices and settle plates at three locations, head of bed/chair two feet away from patient head, foot of bed/chair eight feet away from head, and at the exit of the patient room.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this observational study is to describe the environmental aerosolization patterns burden of RSV in the air and on surfaces in surrounding adult patients in a real-life setting. Specific objectives are to determine the particle size distribution and the quantity of airborne pathogens dispersed by symptomatic participants, to establish a spatial model of airborne emission and subsequent surface burden of RSV emission and dispersal in clinical settings (emergency department and inpatient units; 1 foot vs. 3-6 feet vs. 8-10 feet), and to obtain information regarding the potential association of illness severity and risk factors to the scale of airborne dispersal (e.g., super spreaders). This study will be used to collect data of the emission patterns of RSV. Subsequent investigations will help guide policymakers in the assessment of the airborne exposure risk to RSV and the implementation of appropriate infection prevent measures such as respirators and face masks.

The investigators hypothesize that the airborne emission patterns of Respiratory Syncytial Virus varies between individual patients. The investigators are proposing to assess the particle size and spatial distribution of airborne RSV emitted by affected patients within a routine care environment:

1. Characterize individuals who develop respiratory illnesses caused by RSV in terms of demographics, co-morbid conditions, prior vaccinations (e.g., influenza vaccine, DTAP), use of antivirals, and severity of illness (fever, respiratory symptoms, malaise).
2. Determine the particle size distribution patterns and quantities of the pathogen in two settings, an emergency department and an inpatient unit (ICU and non-ICU settings).
3. Establish a spatial model (1 foot vs. 3-6 feet vs. 8-10 feet) of airborne pathogen dispersal and subsequent surface burden in two settings, an emergency department and an inpatient unit (ICU and non-ICU settings).
4. Determine the correlation between the human aerosolization patterns and the severity of illness (fever, respiratory symptoms, malaise) in individual participants (super spreader?).

DETAILED DESCRIPTION:
Research Design and Methods The main objective of this study is to identify and determine airborne emission and subsequent surface burden patterns of RSV in naturally infected patients.

Patient Information:

Patients seen at the Emergency Department( ED) or admitted to the hospital with respiratory symptoms and diagnosed with RSV are eligible for enrollment. The results of routine in-house laboratory diagnostic tests such as the Respiratory Viral Panel (RVP) will be used to identify patients.

Setting:

Wake forest baptist medical center (WFBMC) is an 885 bed tertiary care teaching hospital. There are approximately 36,000 inpatient admissions and >89,000 ED visits annually (pediatric/adult). Air sampling is conducted in patient rooms under turbulent airflows (6 total air changes/hour) at approximately 20°C temperature and 40% Relative Humidity. Air is filtered by ANSI/ASHRAE 52.2 compliant endfilters with a minimum efficiency reporting value of 15.

Sampling:

One nasopharyngeal swab will be obtained from each subject. The sample will be used to confirm RSV infection and determine the amount of the pathogen carried by the individual. Samples will be inoculated into Becton Dickinson Universal Viral Transport System (VTM, BD Diagnostics, Franklin Lakes, NJ) for real-time reverse transcriptase PCR (rRT-PCR) analysis.

One-time air samples will be collected using six-stage Andersen air sampling devices and settle plates at three locations, head of bed/chair two feet away from patient head, foot of bed/chair eight feet away from head, and at the exit of the patient room (11):

Samples will be collected in viral transport media (VTM), supplemented with RNA stabilization buffer (Qiagen AVL buffer) and carrier RNA and then stored at -80C. Carrier RNA will serve as both a carrier and an internal control by containing genomic RNA of the plant tobacco mosaic virus. A 540 ul volume of RNA sample will be purified with the QIAmp Viral RNA Mini Extraction Kit and concentrated approximately 10-fold. RSV serotypes A and B as well as the control viral tobacco mosaic virus RNA will be detected by reverse transcription and quantitative PCR. Additionally, nNasopharyngeal swab with also be used for cultures with inoculation in petri dish containing RSV specific media.

The surface burden of RSV will be assessed by placement of open standard Petri dishes filled with VTM at the three air sampling locations. The covers of the Petri dishes will be removed at the beginning of and closed after the air sampling session. Selected environmental surfaces will be sampled with sterile swabs moistened with VTM or TSB broth. A two square inch area will be swabbed once at three high-touch locations daily: head of the bed hand rail, middle of food tray table, and a table/horizontal surface at back of room (approximately 10 feet away past foot of bed). The swabs will be vortexed for 30 seconds, and processed as described for RSV detection in air samples.

During the sampling health care professional (HCP) and study staff will wear respirators (N-95) to reduce the risk of external contamination due to potential RSV carrier status. The respirators will be collected and a two square inch midsection of the respirator will be cut out using sterile scissors. The cut-outs are placed in 2mLs VTM or TSB broth and frozen. After thawing, samples are vortexed/agitated, and further processed as described for the RSV samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients > age 18, seen at the Emergency Department or admitted to the hospital with respiratory symptoms and diagnosed with RSV infection

Exclusion Criteria:

* less than age 18
* Mechanically intubated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at the Emergency Department or admitted to the hospital with respiratory symptoms and diagnosed with RSV are eligible for enrollment. The results of routine in-house laboratory diagnostic tests such as the Respiratory Viral Panel (RVP) will be used to identify patients.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
airborne emission patterns of Respiratory Syncytial Virus | 30min - 1 hour
  Determine the particle size distribution patterns and quantities of RSV pathogen, establish a spatial model (1 foot vs. 3-6 feet vs. 8-10 feet) of airborne pathogen dispersal and subsequent surface burden in two settings, an emergency department and an inpatient unit (ICU and non-ICU settings)

SECONDARY OUTCOMES:
Risk of RSV infection based on emission pattern | 72 hours
  Determine the correlation between the human aerosolization patterns and the severity of illness (fever, respiratory symptoms, malaise) in individual participants (super spreader?).

CONTACTS AND LOCATIONS:
Overall Officials: Werner Bischoff, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No